CLINICAL TRIAL: NCT03840681
Title: Assessment of Guided Bone Regeneration in Atrophic Anterior Maxilla Using Native Collagen vs Titanium Reinforced Polytetraflouroethelene Membranes Using an Organic Bovine Bone Mineral
Brief Title: Assessment of Guided Bone Regeneration in Atrophic Anterior Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohab Fathy Metwally, Master student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMetwally
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Guided Bone Regeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Each patient will be given a code by the researcher ( T.A ) and the observer will be blind to which group this case belongs Patients,evaluators and statistican will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ridge augmentation by collagen membrane (Experimental): * Intra operative procedures (for both groups) followed by CBCT will be taken for every patient.
  * Local anesthesia will be given to the patient.
  * Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
  * Flap will be done.
  * bone decortication will be done using surgical round bur, anorganic bovine bone derived mineral will be packed at defected area then covered at the defected area by a collagen membrane which will be stabilized by tacks.
  * The site will then be copiously irrigated with saline in preparation for closure.
  * The flap will then be closed using interrupted 4/0 resorbable sutures.
  Interventions: Other: Augmentation
- augmentation by titanium reinforced PTFE (Active Comparator): * Intra operative procedures (for both groups) followed by CBCT will be taken for every patient.
  * Local anesthesia will be given to the patient.
  * Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
  * Flap will be done.
  * bone decortication will be done using surgical round bur, anorganic bovine bone derived mineral will be packed at the defected area then covered by a titanium reinforced polytetraflouroethelene membrane which will be stabilized by tacks.
  * The site will then be copiously irrigated with saline in preparation for closure.
  * The flap will then be closed using interrupted 4/0 resorbable sutures.
  Interventions: Other: Augmentation

INTERVENTIONS:
Other: Augmentation — non invasive technique to increase bone width and eliminate need for second surgery

SUMMARY:
Guided bone regeneration (GBR) is a surgical technique that uses barrier membranes to promote osteoblast cells proliferation and exclude other cells such as epithelium and connective tissue cells. GBR is often combined with bone grafting procedures.

Using Absorbable membranes like collagen membrane will reduce treatment time by decreasing need for second surgery

DETAILED DESCRIPTION:
Assessment of Guided Bone Regeneration in Atrophic Anterior Maxilla using native Collagen vs Titanium Reinforced Polytetraflouroethelene Membranes using an organic bovine Bone mineral.Reconstructive surgery is necessary before implant placement to regenerate bone defects caused by atrophy, dental trauma, extractions or periodontal disease . Success rate of implants is related to the correct position and angulation of implants in residual crest, so that height and thickness of bone augmentation can allow predictable results ,With this in mind, it is important to establish sound clinical concepts with clearly defined parameters that lead to successful esthetics in the anterior maxilla, with long-term stability of the peri-implant tissues.

The most popular surgical procedures to obtain bone augmentation are: bone grafts, guided bone regeneration, maxillary sinus floor elevation, and bone osteogenesis distraction.

Guided bone regeneration (GBR) is a surgical technique that uses barrier membranes to promote osteoblast cells proliferation and exclude other cells such as epithelium and connective tissue cells. GBR is often combined with bone grafting procedures.

Bone grafts are integrated into native bone with three different processes: osteogenesis, osteoinduction and osteoconduction; Osteogenesis is the formation of new bone from osteocompetent cells and is the only process where the graft itself can induce Bone augmentation, Osteoinduction induces Bone Augmentation from the differentiation and stimulation of mesenchymal cells by the bone-inductive proteins, Osteoconduction is the formation of Bone Augmentation along a scaffold from osteocompetent cells of the recipient site .

There are 2 Types of membranes:

III. Non Resorbable membrane IV. Resorbable membrane

Non-resorbable membranes:

With the presentation of the ﬁrst successful GBR procedures and the subsequent wide and successful application of ePTFE membranes, this material became a standard for bone regeneration. Expanded PTFE is characterized as a polymer with high stability in biological systems. It resists breakdown by host tissues and by microbes and does not elicit immunologic reactions. A frequent complication with membrane application in conjunction with implants is membrane exposure and infection Wound dehiscence and membrane exposure have been reported to impair the amount of bone regenerated in a number of experimental animal and clinical investigations

Bioresorbable membranes:

The requirement of second surgical procedure for the removal of Non Resorbable barrier membrane(NRBM) led to the introduction of bioresorbable barrier membranes (RBM). The advantages of RBM compared to NRBM were as follows:

1. Improved soft tissue healing,
2. Incorporation of the membranes by the host tissues (depending on material properties),
3. Quick resorption in case of exposure, eliminating bacterial contamination. Today, a lot of RBM are commercially available including collagen, freeze-dried fascia lata, freeze-dried dura mater allografts, polyglactin-acid, polylactic acid, polyglycolic acid, polyorthoester, polyurethane, polyhydroxybutyrate, etc.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with atrophied anterior maxillary ridge area.

  * Age: 18 years and older.
  * No intraoral soft and hard tissue pathology.
  * No systemic condition that contraindicate bone augmentation

Exclusion Criteria:

* Heavy smokers more than 20 cigarettes per day.(32)
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems.
* Disorders to bone augmentation are related to history of radiation therapy to the head and neck neoplasia.
* Pregnant or nursing women.
* Patients with uncontrolled diabetes mellitus, rheumatoid arthritis or osteoporosis.
* Patient with previous history of radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Height and width of bone gained | After 6 monthes
  Height and width of bone gained will be measured from CBCT
Bone area percentage | After 6 monthes
  Bone area percentage will be measured by Histo-morphometric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed m Atef, Principal Investigator — Cairo U

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lopez MA, Andreasi Bassi M, Confalone L, Carinci F. REGENERATION OF ATROPHIC CRESTAL RIDGES WITH RESORBABLE LAMINA: TECHNICAL NOTE. J Biol Regul Homeost Agents. 2015 Jul-Sep;29(3 Suppl 1):97-100. PMID 26511187
- [Background] Esposito M, Grusovin MG, Coulthard P, Worthington HV. The efficacy of various bone augmentation procedures for dental implants: a Cochrane systematic review of randomized controlled clinical trials. Int J Oral Maxillofac Implants. 2006 Sep-Oct;21(5):696-710. PMID 17066630
- [Background] Sorni M, Guarinos J, Garcia O, Penarrocha M. Implant rehabilitation of the atrophic upper jaw: a review of the literature since 1999. Med Oral Patol Oral Cir Bucal. 2005 Apr 1;10 Suppl 1:E45-56. English, Spanish. PMID 15800467
- [Background] Hoexter DL. Bone regeneration graft materials. J Oral Implantol. 2002;28(6):290-4. doi: 10.1563/1548-1336(2002)0282.3.CO;2. PMID 12498538
- [Background] Chiapasco M, Zaniboni M, Boisco M. Augmentation procedures for the rehabilitation of deficient edentulous ridges with oral implants. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:136-59. doi: 10.1111/j.1600-0501.2006.01357.x. PMID 16968389
- [Background] Karring T, Cortellini P, Lindhe J. Regenerative periodontal therapy. In: Lindhe J, Karring T, Lang NP, editors. Clinical periodontology and implant dentistry. Copenhagen: Munksgaard, 1997: 597-646.
- [Background] Schliephake H, Kracht D. Vertical ridge augmentation using polylactic membranes in conjunction with immediate implants in periodontally compromised extraction sites: an experimental study in dogs. Int J Oral Maxillofac Implants. 1997 May-Jun;12(3):325-34. PMID 9197097
- [Background] Gotfredsen K, Nimb L, Buser D, Hjorting-Hansen E. Evaluation of guided bone generation around implants placed into fresh extraction sockets: an experimental study in dogs. J Oral Maxillofac Surg. 1993 Aug;51(8):879-84; discussion 885-6. doi: 10.1016/s0278-2391(10)80108-9. PMID 8336225
- [Background] Kohal RJ, Trejo PM, Wirsching C, Hurzeler MB, Caffesse RG. Comparison of bioabsorbable and bioinert membranes for guided bone regeneration around non-submerged implants. An experimental study in the mongrel dog. Clin Oral Implants Res. 1999 Jun;10(3):226-37. doi: 10.1034/j.1600-0501.1999.100306.x. PMID 10522183
- [Background] Becker W, Dahlin C, Becker BE, Lekholm U, van Steenberghe D, Higuchi K, Kultje C. The use of e-PTFE barrier membranes for bone promotion around titanium implants placed into extraction sockets: a prospective multicenter study. Int J Oral Maxillofac Implants. 1994 Jan-Feb;9(1):31-40. PMID 8150510
- [Background] Gher ME, Quintero G, Assad D, Monaco E, Richardson AC. Bone grafting and guided bone regeneration for immediate dental implants in humans. J Periodontol. 1994 Sep;65(9):881-91. doi: 10.1902/jop.1994.65.9.881. PMID 7990026
- [Background] Elgali I, Omar O, Dahlin C, Thomsen P. Guided bone regeneration: materials and biological mechanisms revisited. Eur J Oral Sci. 2017 Oct;125(5):315-337. doi: 10.1111/eos.12364. Epub 2017 Aug 19. PMID 28833567
- [Background] McAllister BS, Haghighat K. Bone augmentation techniques. J Periodontol. 2007 Mar;78(3):377-96. doi: 10.1902/jop.2007.060048. PMID 17335361
- [Background] Hutmacher D, Hurzeler MB, Schliephake H. A review of material properties of biodegradable and bioresorbable polymers and devices for GTR and GBR applications. Int J Oral Maxillofac Implants. 1996 Sep-Oct;11(5):667-78. PMID 8908867